CLINICAL TRIAL: NCT02181608
Title: Traits Associated With Early Life Stress Among Treatment-Seeking Alcoholics
Status: Withdrawn | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140137; 14-AA-0137
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2015-03-24

CONDITIONS: Fear; Stress; Alcohol Dependence
Keywords: Alcohol Dependence; Fear Conditioning; Stress; Alcohol
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Researchers want to see if people with alcohol dependence have more trouble learning to feel calm, or learn to fear things more easily, than non-alcoholics and to study how early life stress (ELS) affects these things.

Objective:

- To see if people with alcohol dependence and/or ELS have a harder time learning to feel calm than people without these conditions.

Eligibility:

* Adults age 21 65 with diagnosed alcohol dependence, with/without ELS.
* Healthy volunteers age 21 65 with/without ELS.

Design:

* All participants will be screened with medical history and physical exam. They will have blood and urine tests, and a psychological assessment.
* Participants with alcohol dependence will:
* be at the NIH Clinical Center for 4 weeks. Then they will have weekly telephone calls and 3 in-person visits over 3 months.
* follow the NIH alcohol treatment program during the study. They cannot take psychiatric medications.
* rate their alcohol craving, depression, and anxiety throughout the study.
* have fear conditioning and extinction sessions that use noise and mild electric shock. Some take place during a functional MRI (fMRI) scan. Participants will lie in a machine that takes images, while they perform tasks.
* listen to recordings that describe stressful events. They will rate their feelings and have blood drawn through an intravenous (IV) line.
* have their hormone response to stress tested. They will take a pill and get a hormone via an IV, then have blood drawn.
* Healthy volunteers will:
* have 2 inpatient stays, each lasting a few days. They will answer questions about how they feel.
* have fear conditioning and extinction sessions, including fMRI.
* have blood drawn several times.

DETAILED DESCRIPTION:
Objective:

The primary objective of the study is to evaluate the role of early life stress (ELS), alcohol dependence (AD), and their interaction in psychophysiology and neural mechanisms of fear conditioning and extinction.

The main outcome of interest is fear extinction, as measured by laboratory-based and fMRI paradigms. Secondary objectives of the study include: (1) explore the impact of early life stress on behavioral and endocrine response to challenge procedures among individuals with AD; (2) explore differences in reward processing, emotion processing, and neural response to alcohol beverages as measured by fMRI as a function of AD and ELS; and (3) examine the relationship between fear extinction and clinical outcomes in our patient sample.

Study Population:

The study sample includes four groups: 1) treatment-seeking individuals with alcohol dependence (AD) and ELS exposure; 2) treatment seeking individuals with alcohol dependence without ELS exposure; 3) healthy social drinkers without alcohol use disorders (AUD) but with ELS exposure; and 4) healthy social drinkers without AUD and without ELS exposure. Target accrual for each of these groups is 25.

Design:

All participants will be evaluated for fear conditioning and extinction using two separate paradigms: an out-of-the scanner shock conditioning extinction procedure that utilizes acoustic startle, and a shock conditioning extinction procedure combined with fMR imaging that utilizes galvanic skin response. In addition, the two alcohol dependent groups will be evaluated for several biomarkers including a guided imagery procedure designed to induce stress and/or craving for alcohol, and an assessment of hypothalamic-pituitary-adrenal (HPA) axis function.

Outcome Measures:

Primary outcome measures include fear-potentiated startle responses and galvanic skin responses; and neural BOLD fMRI responses during presentation of fear associated stimuli. Secondary and exploratory measures in alcohol dependent subjects include measures of distress and craving for alcohol in response to guided imagery scripts; neuroendocrine stress responses and clinical outcomes (alcohol consumption and self-reported anxiety and mood symptoms).

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for AD+/ELS+ group:

* Between 21 and 65 years of age
* Ability to provide written informed consent as determined by successful completion of consent quiz prior to signing consent
* Females: Negative urine pregnancy test, not currently breastfeeding
* Diagnosed with alcohol dependence according to Diagnostic and Statistical Manual for Mental Disorders-Fourth Edition (DSM IV)
* Alcohol consumption within the past month provided by self-report
* Specify alcohol as their preferred drug in a clinical interview
* Minimum score of moderate level of exposure for at least two categories of ELS or score of severe level of exposure for at least on category of ELS as measured by the CTQ (categories include: physical, sexual, and emotional abuse; and physical and emotional neglect; severity level varies by category, and is standardized by the creators of the CTQ)

Inclusion criteria for AD+/ELS- group:

* Between 21 and 65 years of age
* Ability to provide written informed consent as determined by successful completion of consent quiz prior to signing consent
* Females: Negative urine pregnancy test, not currently breastfeeding
* Diagnosed with alcohol dependence according to DSM IV
* Alcohol consumption within the past month provided by self-report
* Specify alcohol as their preferred drug in a clinical interview

Inclusion criteria for AD-/ELS+ group:

* Between 21 and 65 years of age
* Ability to provide written informed consent as determined by successful completion of consent quiz prior to signing consent
* Females: Negative urine pregnancy test, not currently breastfeeding
* Minimum score of moderate level of exposure for at least two categories of ELS or score of severe level of exposure for at least on category of ELS as measured by the CTQ (categories include: physical, sexual, and emotional abuse; and physical and emotional neglect; severity level varies by category, and is standardized by the creators of the CTQ)

Inclusion criteria for AD-/ELS- group:

* Between 21 and 65 years of age
* Ability to provide written informed consent as determined by successful completion of consent quiz prior to signing consent
* Females: Negative urine pregnancy test, not currently breastfeeding

EXCLUSION CRITERIA:

Exclusion criteria for AD+/ELS+ group:

* Neurological symptoms of the wrist or arm, e.g., carpal tunnel syndrome, as determined by history and physical exam
* Chronic use of psychotropic medications within four weeks of the study, with the exception of fluoxetine, for which the exclusionary time period is six weeks. Incidental use of psychotropic medications is allowed but any use must be discontinued prior to the study for a time period exceeding 5 half-lives of the medication in question.
* Presence of any current or past DSM IV diagnosis of bipolar disorder, or psychotic disorder (e.g, schizophrenia, schizoaffective disorder), or substance dependence other than alcohol, nicotine, or caffeine.
* Major medical problems (e.g., central nervous system (CNS), cardiovascular, respiratory, gastrointestinal (GI), hepatic, renal, endocrine, reproductive) that in the judgment of the MAI, in consultation with relevant Clinical Center consult services, cannot be adequately managed at the Clinical Center
* Presence of ferromagnetic objects in the body, fear of enclosed spaces, or other standard contraindication to MRI, as determined by self-report
* Left-handedness

Exclusion criteria for AD+/ELS- group:

* Neurological symptoms of the wrist or arm, e.g., carpal tunnel syndrome, as determined by history and physical exam
* Chronic use of psychotropic medications within four weeks of the study, with the exception of fluoxetine, for which the exclusionary time period is six weeks. Incidental use of psychotropic medications is allowed but any use must be discontinued prior to the study for a time period exceeding 5 half-lives of the medication in question.
* Presence of any current or past DSM IV diagnosis of bipolar disorder, or psychotic disorder (e.g, schizophrenia, schizoaffective disorder), or substance dependence other than alcohol, nicotine, or caffeine.
* Major medical problems (e.g., CNS, cardiovascular, respiratory, GI, hepatic, renal, endocrine, reproductive) that in the judgment of the MAI, in consultation with relevant Clinical Center consult services, cannot be adequately managed at the Clinical Center
* Presence of ferromagnetic objects in the body, fear of enclosed spaces, or other standard contraindication to MRI, as determined by self-report

Score above minimal for one or more categories of ELS as measured by the CTQ

-Left-handedness

Exclusion criteria for AD-/ELS+ group:

* Neurological symptoms of the wrist or arm, e.g., carpal tunnel syndrome, as determined by history and physical exam
* Chronic use of psychotropic medications within four weeks of the study, with the exception of fluoxetine, for which the exclusionary time period is six weeks. Incidental use of psychotropic medications is allowed but any use must be discontinued prior to the study for a time period exceeding 5 half-lives of the medication in question.
* Presence of any current or past DSM IV diagnosis of bipolar disorder, or psychotic disorder (e.g, schizophrenia, schizoaffective disorder), or substance dependence other than alcohol, nicotine, or caffeine.
* Major medical problems (e.g., CNS, cardiovascular, respiratory, GI, hepatic, renal, endocrine, reproductive) that in the judgment of the MAI, in consultation with relevant Clinical Center consult services, cannot be adequately managed at the Clinical Center
* Presence of ferromagnetic objects in the body, fear of enclosed spaces, or other standard contraindication to MRI, as determined by self-report
* Current or past DSM IV diagnosis of alcohol dependence or abuse
* Currently seeking treatment for alcohol problems as assessed by self-report
* Positive urine drug test at screening (for opiates, cannabinoids, amphetamines, cocaine, benzodiazepines)
* Positive breathalyzer test at screening
* Alcohol abstainer
* Left-handedness

Exclusion criteria for AD-/ELS- group:

* Neurological symptoms of the wrist or arm, e.g., carpal tunnel syndrome, as determined by history and physical exam
* Chronic use of psychotropic medications within four weeks of the study, with the exception of fluoxetine, for which the exclusionary time period is six weeks. Incidental use of psychotropic medications is allowed but any use must be discontinued prior to the study for a time period exceeding 5 half-lives of the medication in question.
* Presence of any current or past DSM IV diagnosis of bipolar disorder, or psychotic disorder (e.g, schizophrenia, schizoaffective disorder), or substance dependence other than alcohol, nicotine, or caffeine.
* Major medical problems (e.g., CNS, cardiovascular, respiratory, GI, hepatic, renal, endocrine, reproductive) that in the judgment of the MAI, in consultation with relevant Clinical Center consult services, cannot be adequately managed at the Clinical Center
* Presence of ferromagnetic objects in the body, fear of enclosed spaces, or other standard contraindication to MRI, as determined by self-report
* Score above minimal for one or more categories of ELS as measured by the CTQ
* Current or past DSM IV diagnosis of alcohol dependence or abuse
* Currently seeking treatment for alcohol problems as assessed by self-report
* Positive urine drug test at screening (for opiates, cannabinoids, amphetamines, cocaine, benzodiazepines)
* Positive breathalyzer test at screening
* Alcohol abstainer
* Left-handedness

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06-19; Primary Completion 2015-03-24 (Actual); Study Completion 2015-03-24 (Actual)

PRIMARY OUTCOMES:
To compare physiological and neural outcomes in treatment-seeking alcoholics across multiple challenge procedures as a function of early life stress (ELS) exposure. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)

REFERENCES:
- [Background] Heilig M, Thorsell A, Sommer WH, Hansson AC, Ramchandani VA, George DT, Hommer D, Barr CS. Translating the neuroscience of alcoholism into clinical treatments: from blocking the buzz to curing the blues. Neurosci Biobehav Rev. 2010 Nov;35(2):334-44. doi: 10.1016/j.neubiorev.2009.11.018. Epub 2009 Nov 24. PMID 19941895
- [Background] Prescott CA, Kendler KS. Genetic and environmental contributions to alcohol abuse and dependence in a population-based sample of male twins. Am J Psychiatry. 1999 Jan;156(1):34-40. doi: 10.1176/ajp.156.1.34. PMID 9892295
- [Background] Chartier KG, Hesselbrock MN, Hesselbrock VM. Development and vulnerability factors in adolescent alcohol use. Child Adolesc Psychiatr Clin N Am. 2010 Jul;19(3):493-504. doi: 10.1016/j.chc.2010.03.004. PMID 20682217